CLINICAL TRIAL: NCT00599261
Title: Impact of Pocket Revision on the Rate of Infection and Other Complications in Patients Requiring Pocket Manipulation for Generator Replacement and/or Lead Replacement or Revision: A Prospective Randomized Study
Brief Title: MAKE IT CLEAN, Impact of Pocket Revision on the Rate of Infection and Other Complications in Patients Requiring Pocket Manipulation for Generator Replacement and/or Lead Replacement or Revision: A Prospective Randomized Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Associate Professor of Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10995
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Infection
Keywords: Cardiac Pacemaker, Artificial
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Removal of the fibrotic pocket surrounding the generator and leads
  Interventions: Procedure: ICD/pacemaker pocket revision
- 2 (Experimental): Tissue is not removed
  Interventions: Procedure: ICD/pacemaker pocket revision

INTERVENTIONS:
Procedure: ICD/pacemaker pocket revision — Pocket revision consists of complete removal of the fibrous capsule surrounding the device and leads

SUMMARY:
To determine the effect of scar tissue removal on the rate of infection and any other complications such as bleeding in patients with an ICD or pacemaker who have the device generator or leads replaced or repositioned.

DETAILED DESCRIPTION:
This is a randomized, prospective, single-blind study that evaluates the effect of removal of scar tissue during pacemaker/ICD pocket revision on infection and complications. Subjects will be randomly assigned to either removal of the scar tissue surrounding the implanted device during device replacement or to device replacement without removal of this tissue. Subjects will be followed for one year post-procedure for the occurrence of infection, bleeding/hematoma, or other complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater
2. Willingness to provide written informed consent
3. Subjects presenting for any of the following:

   1. pacemaker/ICD generator change
   2. pacemaker/ICD lead replacement
   3. pacemaker/ICD lead revision
   4. pacemaker/ICD upgrades

Exclusion Criteria:

1. Age less than 18 years
2. Unwillingness to provide written informed consent
3. Subjects unable to give consent
4. Pregnant or nursing women
5. Patients who have undergone pocket revision or manipulation less than 365 days prior
6. Patients who have undergone pacemaker or ICD implantation less than 365 days prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Oral temperature, edema/redness/drainage and/or severity of pain at incision site, presence of chills, reported fever | 1 year

SECONDARY OUTCOMES:
If primary outcome measures are positive, blood and/or device cultures and lab work may be obtained | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Hospital, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Lakkireddy D, Pillarisetti J, Atkins D, Biria M, Reddy M, Murray C, Bommana S, Shanberg D, Adabala N, Pimentel R, Dendi R, Emert M, Vacek J, Dawn B, Berenbom L. IMpact of pocKet rEvision on the rate of InfecTion and other CompLications in patients rEquiring pocket mAnipulation for generator replacement and/or lead replacement or revisioN (MAKE IT CLEAN): A prospective randomized study. Heart Rhythm. 2015 May;12(5):950-6. doi: 10.1016/j.hrthm.2015.01.035. Epub 2015 Jan 24. PMID 25625720